CLINICAL TRIAL: NCT03534271
Title: The Accuracy of Smartphone Pulse Oximetry in Patients Visiting an Outpatient Pulmonary Function Lab for a 6-Minute Walk Test
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brady Scott, Assistant Professor, Director of Clinical Education, Rush University Medical Center
Other Study IDs: 18022702
Record Dates: First submitted 2018-05-08; First posted 2018-05-23 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: iPhone with Kenek Edge and Samsung S8 — Smartphones with pulse oximetry and heart rate monitoring capabilities

SUMMARY:
The primary aim of this research is to determine the accuracy of smartphone pulse oximeters in detecting blood oxygen saturations, episodes of desaturations, and heart rate by comparing results to a Masimo© hospital-grade pulse oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* 18 years and older
* Visiting the pulmonary function laboratory at Rush University Medical Center for a 6-minute walk test that agree to participate.

Exclusion Criteria:

* Under the age of 18 years
* High blood pressure above 180/90 mm Hg or pressure below 70/50 mm Hg
* Dizzy, lightheaded or have severe headaches at time of enrollment
* SpO2 at or below 85% on supplemental oxygen
* On oxygen greater than 4 liters per minute
* Gait issues that may result in a fall or patient walks with a walker and did not bring the device to this visit

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients visiting a pulmonary function lab for 6-minute walk test
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Modi AM, Kiourkas RD, Li J, Scott JB. Reliability of Smartphone Pulse Oximetry in Subjects at Risk for Hypoxemia. Respir Care. 2021 Mar;66(3):384-390. doi: 10.4187/respcare.07670. Epub 2020 Oct 6. PMID 33023999

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 47 subjects that started the study, completed the study
Groups:
- Six Minute Walk Group: Patients undergoing six minute walk
Period: Overall Study
Arm/Group | Six Minute Walk Group
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Six Minute Walk Group: Patients undergoing a six minute walk
Arm/Group | Six Minute Walk Group
Number analyzed (Participants) | 47
Age, Customized [Number; unit: years]
  Age >=18 years | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Black/African American | NA — not analyzed
  White/Caucasian | NA — not analyzed
  Hispanic/Latinx | NA — not analyzed
  Asian | NA — not analyzed
Region of Enrollment [Number; unit: participants]
  United States | 47
Age [Median (Inter-Quartile Range); unit: years] | 69 [57 to 76]

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Smartphone Pulse Oximeters
Description: Accuracy of smartphone pulse oximeter after 6 minute walk Posttest SpO2 %
Time Frame: immediately after the 6 minute walk test
Population: all participants
Measure: Median (Inter-Quartile Range); unit: percentage of oxygen saturation
Groups:
- All Subjects: Subjects doing a six minute walk test
Arm/Group | All Subjects
Number analyzed (Participants) | 47
percentage of oxygen saturation | 98 [96 to 99]

ADVERSE EVENTS:
Time Frame: While each subject participated in the study. No follow up was made.
Description: 47 patient started and completed the study
Groups:
- Six Minute Walk Group: Subjects participating in six minute walk
Arm/Group | Six Minute Walk Group
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03534271/Prot_SAP_000.pdf